CLINICAL TRIAL: NCT04758351
Title: Prospective Study on the Evaluation, Patient Reported Outcomes and Effectiveness of Treatment for Chronic Cough in Secondary Care
Brief Title: Prospective Study on the Evaluation, Patient Reported Outcomes and Effectiveness of Treatment for Chronic Cough
Acronym: PROCOUGH
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Collaborators: Merck Canada Inc. (Industry); University of Manchester (Other); University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: 59689
Record Dates: First submitted 2021-02-05; First posted 2021-02-17 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2024-09

CONDITIONS: Chronic Cough
Keywords: Evaluation; Patient reported; Effectiveness; Treatment; Secondary Care
MeSH Terms: conditions — Chronic Cough

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Remaining cells and supernatant from sputum processing will be stored and used to analyze neuro-inflammatory cytokines and protein biomarkers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases - Patients with chronic cough: Patients referred to secondary care clinic for investigation and treatment for explained chronic cough, refractory chronic cough, and unexplained chronic.
  Interventions: Other: Usual clinical practice

INTERVENTIONS:
Other: Usual clinical practice — Based on European Respiratory Society guidelines on management for chronic cough.

SUMMARY:
Chronic cough is a common troublesome symptom which has a global prevalence of approximately 10%, but with wide variations across continents. The aim of this study is to evaluate the effectiveness of treatment, patient-reported outcomes and burden of disease in patients with chronic cough referred to a specialist clinic. The proposed study will use pre-defined diagnostic criteria, investigations and treatment algorithms such that all recruited patients will undergo the same investigations and follow a set management algorithm. This study will objectively and subjectively assess coughing at baseline and after treatment in a real-world clinical setting. This will allow us to understand the relationship between any objective reduction in cough after treatment, and whether this translates to any significant improvement in subjective questionnaire scores. We will assess the impact of health conditions on lost productivity in monetary units and assess the amount of absenteeism, presenteeism and daily activity impairment attributable to unexplained chronic cough/refractory chronic cough. Finally, a patient survey at the end of the study will evaluate the patients' satisfaction and experience of investigation, management trials and use of questionnaires.

DETAILED DESCRIPTION:
This is a prospective observational single-center study of patients referred to secondary care for investigation and management of explained chronic cough, refractory chronic cough, and unexplained chronic cough. The study will have 4 research visits integrated between standard clinical visits. Patients will be recruited from secondary care clinics. Patient eligibility will be assessed against the study inclusion/exclusion criteria and patients will undergo informed consent in the research centre. Subjects who provide informed consent and are enrolled in the study will undergo screening procedures.

At Visit 1 (screening) data on demographics and medical history will be collected and a complete physical examination will be conducted. Subjects will undergo skin prick testing and spirometry and complete self-reported questionnaires (Leicester Cough Questionnaire, Valuation of Lost Productivity, Work Productivity, Activity, and Impairment, Healthcare Resource Utilization, Reflux Disease Questionnaire, Sino-Nasal Outcome Test, and Global Rating of Change Scale). Subjects will be fitted with a 24-hour cough monitor.

At Visit 2, the 24-hour cough monitor will be removed. Subjects will undergo blood sampling, methacholine challenge, sputum induction, and provide a urine sample.

Between Visits 2 and 3, physicians will provide a single clinical treatment pathway to address the most likely cause of chronic cough. Treatment for chronic cough will be in line with current clinical practice guidelines published by the European Respiratory Society Taskforce on Chronic Cough. Treatment plans will range from 2 weeks to 3 months.

Visit 3 will occur 2 weeks to 3 months following subjects' second clinical visit. Subjects will complete self-reported questionnaires (Leicester Cough Questionnaire, Valuation of Lost Productivity, Work Productivity, Activity, and Impairment, Reflux Disease Questionnaire, Sino-Nasal Outcome Test, and Global Rating of Change Scale) and be fitted with a 24-hour cough monitor.

At Visit 4 the 24-hour cough monitor will be removed. Subjects will undergo blood sampling, sputum induction, and provide a urine sample. Subjects will complete a patient satisfaction survey.

All study procedures will be performed according to local standard operating procedures and be conducted by trained and experienced staff with supervision by medical doctors. Safety will be assessed throughout the study by monitoring for adverse events and serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18-75
2. Patients referred to a specialist primarily with a history of chronic cough (cough lasting >8 weeks)
3. Normal Chest X-ray
4. No Evidence of Airflow Obstruction

Exclusion Criteria:

1. Subjects who are currently established on treatment and their chronic cough is well controlled.
2. Unable to perform acceptable and reproducible spirometry.
3. Current smoker or ex-smoker with ≥20 pack-year smoking history and abstinence of ≤6 months
4. Symptoms of upper respiratory tract infection in the last 1 month which have not resolved
5. Lower respiratory tract infection or pneumonia in the last 1 month
6. Asthma exacerbation in the previous month requiring an increase or start of an inhaled corticosteroid or oral corticosteroid
7. Significant other primary pulmonary disorders in particular; pulmonary embolism, pulmonary hypertension, lung cancer, cystic fibrosis, significant radiologically proven emphysema, interstitial lung disease or bronchiectasis.
8. Any centrally acting medication within the last 2 weeks which in the view of the investigator could influence the coughing. Any participant who is taking amitriptyline, dextromethorphan, pregabalin, gabapentin or opioids will not be eligible to take part in this study unless they are willing and medically able to withdraw from such medication before the start of visit 1. The reason for this is that centrally-acting medications may influence coughing rates at baseline.
9. History of psychiatric illness, drug or alcohol abuse which may interfere in the participation of the trial.
10. Positive Covid-19 test within 2 weeks of screening visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to secondary care for investigation and treatment of explained chronic cough, refractory chronic cough, and unexplained chronic cough.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Changes in objective cough frequency | 3 months
  Change in objective cough frequency pre- and post-treatment among patients referred to secondary care for treatment of explained chronic cough, refractory chronic cough, and unexplained chronic cough.

SECONDARY OUTCOMES:
Correlation in change of objective cough frequency and healthcare utilization | 3 months
  Correlation between pre- and post-treatment change in objective cough frequency and Healthcare Related Utilization among patients referred to secondary care for treatment of explained chronic cough, refractory chronic cough, and unexplained chronic cough. Healthcare utilization is measured by recording the number of visits to family physician, outpatient specialist, number of tests, and medication use.
Correlation in change of objective cough frequency and lost productivity | 3 months
  Correlation between pre- and post-treatment change in objective cough frequency and lost productivity among patients referred to secondary care for treatment of explained chronic cough, refractory chronic cough, and unexplained chronic cough. Lost productivity is measured using the Valuation of Lost Productivity questionnaire which contains a series of questions that evaluate the impact of functional impairment on productivity loss, not just for the individual but also on the work environment.
Correlation in change of objective cough frequency and work productivity and activity | 3 months
  Correlation between pre- and post-treatment change in objective cough frequency and work productivity and activity among patients referred to secondary care for treatment of explained chronic cough, refractory chronic cough, and unexplained chronic cough. Work productivity and activity is measured using the Work Productivity and Activity Impairment Questionnaire which is a 6-item self-administered questionnaire used to assess productivity and impairment because of a specific health problem such as chronic cough.
Correlation in change of quality of life and healthcare utilization | 3 months
  Correlation between pre- and post-treatment change in quality of life and Healthcare Related Utilization among patients referred to secondary care for treatment of explained chronic cough, refractory chronic cough, and unexplained chronic cough. Quality of life is measured using the Leicester Cough Questionnaire. The Leicester Cough Questionnaire is a 7 point Likert scale with a minimum value of 1 indicating chronic cough impacts participant life all of the time and a maximum value of 7 indicating chronic cough impacts participant life none of the time. Healthcare utilization is measured by recording the number of visits to family physician, outpatient specialist, number of tests, and medication use.
Correlation in change of quality of life and lost productivity | 3 months
  Correlation between pre- and post-treatment change in quality of life and lost productivity among patients referred to secondary care for treatment of explained chronic cough, refractory chronic cough, and unexplained chronic cough. Quality of life is measured using the Leicester Cough Questionnaire. The Leicester Cough Questionnaire is a 7 point Likert scale with a minimum value of 1 indicating chronic cough impacts participant life all of the time and a maximum value of 7 indicating chronic cough impacts participant life none of the time. Lost productivity is measured using the Valuation of Lost Productivity questionnaire which contains a series of questions that evaluate the impact of functional impairment on productivity loss, not just for the individual but also on the work environment.
Correlation in change of quality of life and work productivity and activity | 3 months
  Correlation between pre- and post-treatment change in quality of life and work productivity and activity among patients referred to secondary care for treatment of explained chronic cough, refractory chronic cough, and unexplained chronic cough. Quality of life is measured using the Leicester Cough Questionnaire. The Leicester Cough Questionnaire is a 7 point Likert scale with a minimum value of 1 indicating chronic cough impacts participant life all of the time and a maximum value of 7 indicating chronic cough impacts participant life none of the time. Work productivity and activity is measured using the Work Productivity and Activity Impairment Questionnaire which is a 6-item self-administered questionnaire used to assess productivity and impairment because of a specific health problem such as chronic cough.
Patient satisfaction | 3 months
  Patient satisfaction measurements of clinical investigations, treatment, and use of questionnaires among patients referred to secondary care for treatment of explained chronic cough, refractory chronic cough, and unexplained chronic cough. Patient satisfaction will be measured using a 5 point Likert scale where the minimum value is 1 indicating participants were very unsatisfied and the maximum value is 5 indicating participants were very satisfied.
Comparison of change in objective cough frequency and quality of life | 3 months
  Comparison of pre- and post treatment change in objective cough frequency and quality of life among patients referred to secondary care for treatment of explained chronic cough, refractory chronic cough, and unexplained chronic cough. Quality of life is measured using the Leicester Cough Questionnaire. The Leicester Cough Questionnaire is a 7 point Likert scale with a minimum value of 1 indicating chronic cough impacts participant life all of the time and a maximum value of 7 indicating chronic cough impacts participant life none of the time.
Comparison of change in objective cough frequency and participant perceived change in condition | 3 months
  Comparison of pre- and post-treatment change in objective cough frequency and perceived change in condition among patients referred to secondary care for treatment of explained chronic cough, refractory chronic cough, and unexplained chronic cough. Perceived change in condition is measured using the Global Rating of Change Scale which is a 15 value scale. The Global Rating of Change Scale is a 15 point scale with a minimum value of -7 indicating a worse outcome and a maximum value of +7 indicating a better outcome.
Measure the relationship between objective cough frequency and lost productivity | 3 months
  Measure the post treatment relationship between objective cough frequency and lost productivity among patients referred to secondary care for treatment of explained chronic cough, refractory chronic cough, and unexplained chronic cough. Lost productivity is measured using the Valuation of Lost Productivity questionnaire which contains a series of questions that evaluate the impact of functional impairment on productivity loss, not just for the individual but also on the work environment.
Measure the relationship between objective cough frequency and work productivity and activity | 3 months
  Measure the post treatment relationship between objective cough frequency and work productivity and activity among patients referred to secondary care for treatment of explained chronic cough, refractory chronic cough, and unexplained chronic cough. Work productivity and activity is measured using the Work Productivity and Activity Impairment Questionnaire which is a 6-item self-administered questionnaire used to assess productivity and impairment because of a specific health problem such as chronic cough.

OTHER OUTCOMES:
Correlation in exhaled nitric oxide, blood eosinophils, and sputum eosinophils and objective cough frequency and subjective patient reported outcomes | 3 months
  Correlations between exhaled nitric oxide, blood eosinophils, and sputum eosinophils and objective cough frequency and subjective patient reported outcomes pre- and post-treatment in patients referred to secondary care for treatment of explained chronic cough, refractory chronic cough, unexplained chronic cough.
Changes in the quality of life | 3 months
  Changes in the quality of life, measured using the Leicester Cough Questionnaire pre- and post-treatment in patients referred to secondary care for treatment of explained chronic cough, refractory chronic cough, unexplained chronic cough.The Leicester Cough Questionnaire is a 7 point Likert scale with a minimum value of 1 indicating chronic cough impacts participant life all of the time and a maximum value of 7 indicating chronic cough impacts participant life none of the time.
Changes in the perceived disease | 3 months
  Changes in perceived disease improvement, measured using the Global Rating of Change Scale, pre- and post-treatment in patients referred to secondary care for treatment of explained chronic cough, refractory chronic cough, unexplained chronic cough. The Global Rating of Change Scale is a 15 point scale with a minimum value of -7 indicating a worse outcome and a maximum value of +7 indicating a better outcome.
Correlations between improved quality of life and perceived disease improvement | 3 months
  Correlations between improved quality of life, measured using the Leicester Cough Questionnaire, and perceived disease improvement, measure using the Global Rating of Change Scale, pre- and post-treatment in patients referred to secondary care for treatment of explained chronic cough, refractory chronic cough, unexplained chronic cough.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Satia, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- Imran Satia, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Song WJ, Chang YS, Faruqi S, Kim JY, Kang MG, Kim S, Jo EJ, Kim MH, Plevkova J, Park HW, Cho SH, Morice AH. The global epidemiology of chronic cough in adults: a systematic review and meta-analysis. Eur Respir J. 2015 May;45(5):1479-81. doi: 10.1183/09031936.00218714. Epub 2015 Feb 5. No abstract available. PMID 25657027
- [Background] Irwin RS, Baumann MH, Bolser DC, Boulet LP, Braman SS, Brightling CE, Brown KK, Canning BJ, Chang AB, Dicpinigaitis PV, Eccles R, Glomb WB, Goldstein LB, Graham LM, Hargreave FE, Kvale PA, Lewis SZ, McCool FD, McCrory DC, Prakash UBS, Pratter MR, Rosen MJ, Schulman E, Shannon JJ, Hammond CS, Tarlo SM. Diagnosis and management of cough executive summary: ACCP evidence-based clinical practice guidelines. Chest. 2006 Jan;129(1 Suppl):1S-23S. doi: 10.1378/chest.129.1_suppl.1S. No abstract available. PMID 16428686
- [Background] Morice AH, Kastelik JA. Cough. 1: Chronic cough in adults. Thorax. 2003 Oct;58(10):901-7. doi: 10.1136/thorax.58.10.901. PMID 14514949
- [Background] Pratter MR. Overview of common causes of chronic cough: ACCP evidence-based clinical practice guidelines. Chest. 2006 Jan;129(1 Suppl):59S-62S. doi: 10.1378/chest.129.1_suppl.59S. PMID 16428693
- [Background] Sadatsafavi M, Rousseau R, Chen W, Zhang W, Lynd L, FitzGerald JM. The preventable burden of productivity loss due to suboptimal asthma control: a population-based study. Chest. 2014 Apr;145(4):787-793. doi: 10.1378/chest.13-1619. PMID 24337140
- [Background] Andreasson E, Svensson K, Berggren F. PRP11 The validity of the work productivity and activity impairment questionnaire for patients with asthma (WPAIASTHMA): Results from a web-based study. Value in Health. 2003;6(6):780.